CLINICAL TRIAL: NCT00507221
Title: Empiric Therapy of Helminth Co-infection to Reduce HIV-1 Disease Progression
Acronym: THE or PHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Judd Walson, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32274-B; KEMRI SSC #1251; 07-6824-B 01
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: HIV Infections; Helminthiasis
Keywords: HIV; Helminthiasis; Co-infection; Treatment Naive
MeSH Terms: conditions — HIV Infections; Helminthiasis; Coinfection | interventions — Albendazole; Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Arm 1 will receive an intensive regimen of anti-helminthic therapy consisting of albendazole every three months for two years and praziquantel at enrollment and at one year of follow up.
  Interventions: Drug: Albendazole; Drug: Praziquantel
- 2 (Active Comparator): Arm 2 will receive symptomatic diagnosis and treatment of helminth infection as is current standard of care in Kenya.
  Interventions: Drug: Current standard of care in Kenya

INTERVENTIONS:
Drug: Albendazole — Every 3 months for 24 months (enrollment 3, 6, 9, 12, 15, 18, 21, and 24 months):
  400mg/day X 3 days
  Arms: 1
Drug: Praziquantel — At enrollment and 12 months: 25mg/kg X 1
  Arms: 1
Drug: Current standard of care in Kenya — Current standard of care for HIV patients in Kenya based on WHO guidelines.
  Arms: 2

SUMMARY:
Abstract:

Over 25 million HIV-1 infected individuals are currently living in Africa and as many as 50-90% may be co-infected with soil transmitted helminths such as roundworms, hookworms or whipworms. Helminth infection in HIV-1-infected individuals may increase HIV-1 RNA levels and increase the rate of progression of HIV-1 to AIDS. Studies have also shown that successful treatment of helminth co-infection (as documented by clearance of helminth eggs in stool) led to a significant decrease in HIV-1 plasma viral load (-0.36 log10). This change in viral load was significantly greater than that seen in those individuals without documented clearance of their helminth co-infection (+0.67 log10) (p=0.04). Studies conducted in Africa have shown an estimated 2.5-fold increased risk for sexual transmission of the HIV-1 for each log increase in plasma HIV-1 viral load. In addition to direct effects on plasma viral load, the rate of CD4 cell decline in helminth infected individuals may be directly impacted by the significant immune activation seen with such co-infection.

The investigators propose a randomized controlled trial examining the potential benefits of routine empiric helminth eradication in HIV-1 infected adults who do not yet qualify for antiretroviral (ARV) therapy in Kenya. The current standard of care of symptomatic diagnosis and treatment will be compared to a systematic empiric scheduled de-worming program for HIV infected adults. The investigators will compare markers of disease progression including rate of CD4 decline and changes in HIV-1 RNA levels between the two treatment arms.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND: BACKGROUND, SIGNIFICANCE AND RATIONALE

• Epidemiology of HIV-1 and helminth infections in Africa: Over two thirds of all HIV-1 infected individuals live in Africa. An expected 4 million new infections will occur this year in Africa alone. While antiretroviral therapies (ARTs) offer the hope of stemming this tremendous public health disaster, the reality is that many individuals are not able to access ARTs. In addition, millions of HIV infected individuals do not yet qualify for ART based on clinical or immunologic staging criteria. Alternative care strategies to delay immunosuppression and reduce infectivity are critically needed. Treatment of co-infections that are prevalent in areas of high HIV-1 sero-prevalence may be one strategy to address this need.

Helminths represent some of the most common infections of humans throughout the world. It is estimated that over half of all individuals living in Sub-Saharan Africa are infected with at least on species of soil transmitted helminths. Distribution mapping of HIV-1 sero-prevalence and helminth infection prevalence reveal remarkably geographic similarities.

We have recently conducted a large study of helminth infection among HIV-1 infected adults at several sites in Kenya. While rates of helminth co-infection are highest in Kilifi and Nyanza sites, there is a significant rate of co-infection even within the greater Nairobi area.

We also determined that while hookworm was the most common helminth identified in this cohort, the type of helminth infection varied significantly with the location.

• Immunology of helminth co-infection: Helminth infection has been shown to have profound effects on the immune system. Chronic helminth infection leads to a dominant Th2 immune profile, anergy to various antigens, and significant activation of the immune system. These changes suggest that helminth co-infection may significantly affect the host immune response to HIV-1 viral replication and control. Such immune dysregulation may also increase HIV co-receptor expression and result in a cell population more susceptible to HIV infection.

• Th1/Th2 Immune Bias: An important immunologic consequence of helminth infection is the polarization of the immune response to a TH2 subset. This immune modulation by helminth species appears to be important in tempering TH1 cell mediated inflammation and subsequent tissue damage to the host. Such modulation may be detrimental to the HIV-1 infected host by limiting the Th1 immune response that may be important for the control of HIV-1 replication. The TH2/TH1 response to infection is directly influenced by parasite biology. Helminth infection results in specific nematode-elicited macrophages (NeMacs) that directly induce naïve T cells to differentiate into Th2 cells. Cytokine mimics produced by some parasites are also able to directly induce Th2 cells. Other non-protein molecules produced by helminths are able to interact with dendritic cells and induce Th2 cells and Treg cells that produce IL-10 and directly lead to a Th2 shift in naïve T cells.

In addition to being inducers of Th2 cells, there is evidence that helminth infection can directly suppress the Th1 response. This reduction in the Th1 cytokine response is accompanied by a reduction in virus specific CD8+ cytotoxic T lymphocytes (CTL's). Plasma HIV-1 viral load is directly related to HIV-1 specific CTL responses in humans and a reduction in CTL response is associated with a more rapid progression of HIV-1 disease.

• Immune Activation: Individuals residing in Africa display high levels of immune activation. Initial studies of Ethiopian immigrants to Israel revealed elevated levels of plasma IgE and IgG as well as increased levels of eosinophilia that were strongly associated with the presence of helminth infection in this population. These individuals were also found to have significantly activated CD4 lymphocytes that correlated with reduced total CD4 number in this cohort.

Several authors have suggested that this increased activation may be important in the pathogenesis of HIV-1 infection. The uncontrolled T cell destruction characteristic of HIV infection is not due to the direct cytopathic effects of the virus but is more likely the result of activation-induced cell death. Immune activation markers (namely HLA-DR, Ki-67 and CD38) have been shown to be more predictive of CD4 decline than plasma HIV-1 RNA viral load. Treatment of helminth infections can result in reversal of this activated immune state.

Helminth co-infection and clinical HIV-1 disease progression in resource constrained settings • Effect of treatment on HIV-1 RNA: Plasma HIV-1 RNA levels correlate closely with the burden of helminth infection as measured by the number of excreted eggs per gram of stool (p < 0.001). In this same cohort, anti-helminth therapy leading to clearance of helminth eggs in the stool led to a significant decrease in HIV-1 plasma viral load (-0.36 log10) in this cohort. While this effect may appear modest, mathematical modeling suggests that a 0.5 log reduction in HIV-1 RNA levels would slow the onset of AIDS by 3.5 years and would delay the need for antiretroviral medications by almost a full year.

To date, only one randomized controlled trial has been conducted evaluating the effect of treating helminths on markers of HIV-1 progression. In this small unblinded study conducted in Zimbabwe, individuals with schistosomiasis (both with and without HIV-1 infection) were randomized to receive praziquantel at inclusion or after a delay of 3 months. The study found that the HIV-1 infected individuals receiving early treatment of schistosomiasis had no change in plasma HIV-1 RNA levels compared to an increase in HIV-1 RNA levels in the delayed treatment group. However, several other observational studies evaluating the effect of treating helminth co-infection have found that successful eradication of helminths had no effect on plasma HIV-1 RNA levels or even led to transient increases in viral load. We are currently conducting a systematic review for the Cochrane Library evaluating all of the available data examining the effect of treating helminths of HIV-1 RNA levels and CD4 counts.

* Effect of treatment on CD4 count:

Studies evaluating changes in CD4 counts following therapy for helminth co-infection have largely failed to find significant differences. The randomized controlled trial noted above did find that patients treated for helminths in the early treatment group (both HIV seropositive and seronegative) had a increase in absolute CD4 counts compared to no change in CD4 counts in the delayed treatment group (p < 0.05). Another study conducted in Ethiopia found that the treatment of helminth infection in a population of co-infected individuals resulted in a significant increase in absolute CD4 counts (192 versus 279 cells/mm3, p = 0.002). Other studies have shown no significant difference in CD4 decline following anti-helminth treatment. The systematic review currently in preparation has not found a trend towards an effect on CD4 counts in the available studies though all included studies were of short duration (4 months or less).

• Justification of the Study: It is important to determine if empiric deworming can be beneficial for the millions of pre-HAART HIV-1 positive individuals living in helminth endemic areas. Documenting the potential effects of such an intervention on markers of disease progression will serve to inform practical approaches for cost-effective interventions in resource limited settings. Interval anti-helminth therapy may be a feasible option in many areas of the world to delay immunosuppression, to enhance the response to antiretroviral therapy or to reduce infectiousness in HIV-1 infected individuals. In addition, as patients progress to HAART, it is important to determine the ideal timing for helminth eradication.

• Hypothesis: An empiric intensive treatment regimen to eliminate helminths in patients with HIV-1 may impact markers of disease progression, namely CD4 count and plasma HIV-1 RNA levels, when compared to current standard of practice in Kenya.

• Overall General Objectives: To evaluate the effect of an empiric intensive helminth eradication regimen on HIV-1 disease progression in a cohort of HIV-1 infected Kenyan adults who do not meet criteria for highly active antiretroviral therapy.

• Specific Objectives:

1. To evaluate the effect of an intensive, empiric deworming regimen on changes in markers of HIV-1 disease progression, namely time to ART eligibility and time to CD4 count less than 200 and less than 350 cells/mm3 in a cohort of HIV-1 infected adult Kenyans not meeting criteria for antiretrovirals.
2. To determine if intensive treatment of intestinal helminths in HIV-1 infected adults can reduce markers of clinical disease progression as measured by WHO staging criteria, hospitalization and death.

   DESIGNS AND METHODOLOGY • Study Site: The study will be conducted at several HIV care sites in Kenya. The University of Washington has a history of collaborative research with the Kenya Medical Research Institute, the University of Nairobi, and Kenyatta National Hospital; all leading academic institutions in Kenya. Enrollment in the randomized clinical trial will take place at up to three sites in Kenya. The determination of sites will be based on ongoing studies of helminth prevalence in Kenya (Walson JL, Otieno P, ongoing) and may include AMREF/CDC Clinic in Kibera, KNH Comprehensive Care Clinic, KEMRI CCC, Homa Bay District Hospital, Kisii District Hospital, Kisumu District Hospital, Kerugoya District Hospital, Machakos District Hospital, Mbagathi District Hospital, Thika District Hospital, and The Comprehensive Care and Research Clinic at Kilifi District Hospital (CGMR-C).
   * Study Populations:

   Individuals who are 18 years or older, who are not currently on antiretroviral therapy and who are interested in study participation will be enrolled after written informed consent is obtained.

   • Sample Size: Sample size determination - Assuming a power of 90% and alpha of 0.05, we have calculated that 340 individuals would be needed in each arm to detect a difference in CD4 decline of 50 cells/mm3 between the two groups (SD of 200 cells/mm3) over the two years of follow up. Given a maximum expected loss to follow up of approximately 20% over the 24 months of follow up and a maximum of 20% beginning ARV therapy, we will enroll 1200 individuals in the trial to ensure that 340 individuals are available in each arm for analysis. This sample size will also provide greater than 90% power to detect a 0.5 log difference in log10 HIV RNA levels between the treatment arms.
   * Study design:

   Specific Aim 1: randomized clinical trial Specific Aim 2: randomized clinical trial
   * Procedures:

   Summary: We propose a prospective, randomized, controlled trial of an intensive deworming care package versus standard of care in a cohort of HIV-1 seropositive adults who do not yet meet criteria for antiretroviral medications. Participants will be randomized into one of two treatment arms. Arm 1 will receive an intensive regimen of anti-helminthic therapy consisting of albendazole every three months for two years and praziquantel at enrollment and at one year of follow up. Arm 2 will receive symptomatic diagnosis and treatment of helminth infection as is current standard of care in Kenya. The primary objectives of this study are to evaluate changes in CD4 count and HIV-1 RNA over the two years of follow up in each of the study arms.

   Adult men and women participating in or referred to the HIV Care and Treatment Clinics at each of the included sites will be offered screening for eligibility. HIV-1 seropositive individuals with a documented CD4 count greater than 350 cells/mm3 will be considered potentially eligible. Those who agree to participate, are willing and able to provide informed consent, are WHO stage I or II based on clinical exam and history, are 18 years of age or older, have not been treated with worm medication in the previous 4 months and who are not pregnant (based on urine beta-HCG testing if female) will be offered to participate in this trial. Pregnancy testing will be performed at each study visit (every three months) for all premenopausal women. Women who become pregnant during the course of the study will continue to be followed but will not receive any further study medication during pregnancy if they had been randomized to study arm A.
   * Clinical Trial:

   Screening for trial eligibility:

   At each selected clinical trial study site, HIV-1 infected individuals who meet inclusion and exclusion criteria will be informed about the ongoing study. A physical examination will be conducted on all prospective clients, and those found to have clinical pallor or signs of WHO Stage III or IV HIV will be excluded from the study and referred for appropriate medical management. Those who meet criteria and wish to participate will be referred to the study staff for possible enrollment.

   All invited participants will be required to sign written informed consent prior to enrollment. At enrollment, all participants will complete a standardized questionnaire assessing medical and social history and will undergo a complete physical examination. Blood specimens will be collected for full blood count with differential measurement of absolute CD4 count and HIV-1 RNA levels.

   A detailed questionnaire will also be administered in order to assess socio-economic status, living conditions, level of education completed and occupation. This questionnaire will also document potential exposures to helminth infection such as water supply, sanitation facilities, exposure to large bodies of water and type of foot covering used. In addition, a detailed clinical history will also be collected to document any prior illnesses or treatments relevant to HIV-1 or co-infections.

   Detailed information regarding the location of each participant's current residence and any additional residences that they consider as a primary dwelling will also be collected by field workers at each site. Global positioning system information will be collected at the location of each participants site of primary residence to facilitate patient tracing. This information will be stored as well as any other potential contact information available (such as cell phone numbers) in order that participants may be traced for the purposes of the study.

   After signing informed consent and being enrolled, participants will be randomized into one of two treatment arms. The study biostatistician will generate block randomization codes for the sites. Both the investigators and the participants will remain blinded to study arm allocation until randomization occurs.

   All enrolled participants will have scheduled study visits every third month for 24 months (enrollment, months 3, 6, 9, 12, 15, 18, 21 and 24) at the clinic from which they were enrolled. At each follow up visit, a standardized questionnaire designed to assess any change in socio-demographic variables or clinical history will be performed. A physical examination will also be performed at each visit. Blood will be collected at enrollment, months 6, 12, 18 and 24 for measurement of full blood count with differential and CD4 count. Measurement of HIV-1 RNA will be collected at enrollment, the 12 month visit and the 24 month visit. All blood will be separated into plasma and PBMC's (peripheral blood mononuclear cells) and stored for future studies. Any future study utilizing stored specimens will obtain approval from both the Kenya Medical Research Institute and the University of Washington Ethical Review Boards. All participants will provide a single stool sample at the final 24 month follow up visit to determine helminth infection status at that time.

   • Rationale for not screening stool samples at each visit: Participants will not be screened for helminth infection at enrollment or during the course of this study. The only testing for helminth infection status will occur at the final visit. The rationale for this design is principally due to the study objectives. The study is designed to assess the potential benefit of empiric helminth therapy in HIV-1 infected individual's not yet meeting criteria for initiation of antiretroviral medications. As such, it is important to determine if HIV infected individuals in areas of moderate helminth prevalence (20-40%) would benefit from a program of empiric deworming as part of their pre-HAART care package. It is critical that participants be enrolled regardless of helminth infection status in order to determine if empiric therapy should be considered as a useful addition to the care package currently provided to these individuals.

   Storage of stool samples for evaluation of helminth status following completion of the study is also not feasible for several reasons. Most importantly, there are ethical issues related to the collection of samples (and therefore the potential knowledge of infection status) without providing directed therapy. If helminth status is known (or potentially known), the standard of care in Kenya would change from symptomatic screening and treatment to definitive pathogen directed therapy. This would alter the intervention arms in the current study. In addition, the most common helminth at all of the sites sampled in our previous study was hookworm. Hookworm eggs are fragile and rapidly degrade. None of the currently available techniques will preserve hookworm eggs reliably and so any delayed evaluation of helminth infection status is likely to miss many infections and therefore not provide any additional useful information.

   • Laboratory:

   Between ten and twenty millilitres of blood will be drawn each visit where laboratory investigations are being conducted (months 0, 6, 12, 18 and 24). This quantity of blood is being drawn for the following assays:

<!-- -->

1. CD4 measurement (5 mL) will be assessed by FACSCount or FACSCalibur at the individual study sites or at the KEMRI/University of Washington Flow Laboratory at the Centre for Clinical Research in Nairobi, Kenya.
2. Full Blood Counts with Differential (2 mL) will be assessed at each individual study site.
3. Stool microscopy will be performed by technicians with training and certification in the differentiation and quantification of stool helminth species. Stool will be prepared for examination by wet preparation, Kato-Katz technique and formol-ether concentration. Both qualitative and quantitative diagnosis will be made for all helminths identified in stool.
4. Circulating Anodic Antigen (CAA) (3 mL) will be assessed in the Centre for Clinical Research, KEMRI.
5. HIV-1 RNA levels (10 mL) will be quantified at the Kenya Medical Research Institute/Centers for Disease Control, Kenya.

   • Data Management and Analysis: This study is being carried out at several clinical sites in Kenya. Clinical and laboratory data for each participant will be abstracted from routine clinical data forms into standardized trial files. These data will be entered weekly into a computer using a computerized database designed and maintained by the study investigators. Information will be cross checked for accuracy on a bi-weekly basis. All data, both hard and soft copy format, will be stored in locked cabinets with limited access by study staff only. Participants will be identified by a unique study ID number and the code linking the study ID to individual identifying information will be kept in a separate secure location by the principal investigator.

   All data will be collected on preprinted forms and data entered into a software data management program (Teleform SPSS, MS ACCESS or SQL). Data will be collected at enrollment and at each follow up visit on these forms. Following collection, the data forms will be entered into the database as described above. Original data forms will be stored in the study offices with access restricted to study investigators. Following completion of all data collection, the data forms will be archived. At 1-year following completion of the study, identifiers will be removed from the data. Data will be the property or KEMRI and the University of Washington.

   Data verification:

   A data clerk from KEMRI will be employed to hand verify that all data is completed accurately and that the computerized scanned data is comparable to the paper forms. Data will be cleaned by the Principal Investigator, the data manager and data clerk and at that time a second verification of accuracy will be performed.

   Data Analysis:

   Aim 1: All analyses will be intent-to-treat. To assess the success of randomization we will compare baseline characteristics between the 2 randomization groups using Chi-square tests for categorical data and Mann-Whitney U-tests or t-tests for continuous data. To determine the effect of anti-helminth treatment on disease progression markers, we will compare the time to eligibility for ART between the groups and the time to CD4 counts of less than 200 and 350 respectively using Cox regression analysis models. If current treatment guidelines for the initiation of ART change during the course of the study, the analysis plan would incorporate that change in ART eligibility criteria as a date dependent event. In addition, we will compare changes in measurements of mean CD4 count and log10 plasma HIV-1 RNA in the two study arms using linear mixed effects models or linear regression censoring values after initiation of ART.

   Aim 2: To determine the effect of anti-helminth treatment on clinical disease progression markers, we will compare time to changes in WHO Clinical Staging, time to hospitalization, and time to death using Cox regression analysis models. We will also compare the treatment arms for CD4 response to ARVs, and development of IRIS among those who initiate therapy during the course of the trial using regression models.

   Efficacy assessment The primary measure of efficacy for the randomized clinical trial is the time to ART eligibility and the time to CD4 counts of less than 200 and 350 cells/mm3. Secondary measures of efficacy will include changes in WHO Clinical Staging, development of IRIS, time to hospitalization, time to death, time to initiation of ARVs and CD4 response to ARVs as well as the development of IRIS among those who initiate ARVs.

   Safety and loss to follow up All participants will be monitored over the course of the trial for adverse events, laboratory abnormalities and HIV related morbidity. Any participant experiencing National Institutes of Health grade 3-4 toxicity after receipt of anti-helminthic therapy will be withdrawn from the study.

   A Data Safety Monitoring Board (DSMB) will be convened and will meet every 6 months following the start of enrolment to review safety data including all adverse events, protocol violations and any other reported events. In addition, the DSMB will review interim data when 250 patients have completed 12 months of follow up.

   Participants failing to meet a clinic appointment or follow up will be identified and have their study file flagged. If a participant fails to return to clinic within two weeks following a missed appointment, a social worker or peer counselor will attempt to contact the participant to encourage attendance using the contact information provided at enrollment. All attempts at contact will be recorded. If a participant desires to be removed from the study or fails to follow up after 3 consecutive attempts by the peer counselors or social workers to encourage follow up, the participant will be considered lost to follow up. It the study staff is unable to trace the patient for a period of 60 days following a missed appointment, the participant will be considered lost to follow up. If a participant dies in the course of the study, a verbal autopsy will be obtained from family members or household contacts where possible for classification of possible cause of death.

   Participants who meet criteria for the initiation of septrin prophylaxis or ARV's during the course of the study (based on CD4 count or clinical criteria) will be referred for initiation of treatment at the clinic at which they were enrolled. All of the clinics considered as study sites are supported by Government of Kenya and PEPFAR and provide antiretroviral therapy and septrin prophylaxis at no charge to clients who qualify.
   * Time Schedule:

   This study will require approximately 3-4 years for completion. Enrollment will occur over a 6 month period. All participants will be followed for 24 months after enrollment. Thus, it will take approximately 2.5 years to enroll, randomize and complete follow up for all of the patients in the study. An additional 6 months of preparation time will be required to develop the database and prepare each site for study enrollment. Following completion of follow up, we anticipate an additional 6 months will be necessary to complete all laboratory investigations, data analysis, data cleaning and completion of a manuscript.

   • Ethical Considerations:

   • Ethical approval: Study approvals will be obtained from the University of Washington and the KEMRI ethical review boards.

   • Benefits: This study has been designed to address several areas of major public health significance for HIV-1 infected individuals in resource poor settings. If we are able to show that treatment of helminth co-infection in HIV-1 infected individual's delays immunosuppression, millions of HIV infected individuals in resource poor settings may benefit. Participants randomized to the intensive intervention arm will benefit from free treatment and examination given to them. All participants will benefit from intensive clinical and laboratory monitoring.

   • Voluntary Participation: All subjects will provide written informed consent prior to study enrolment. Consent forms will be made available in Swahili as well as in English. All patients will have the opportunity to have the forms explained to them and to ask questions of the investigator prior to study enrollment. Patients will be informed of their right to withdraw consent at any time. Since the participants will spend extra time to participate in the study, they will receive compensation for transport, but no other compensation will be provided to them.

   The field sites where patients will be recruited for screening and enrollment are in Kenya. All of these sites are currently receiving support through CDC Kenya using the PEPFAR mechanism. Laboratory procedures will be performed at each clinic site, in Nairobi and in Seattle, Washington. The study will be reviewed by the Institutional Review Board (IRB) at the University of Washington and the Ethical Review Board (ERC) at the Kenya Medical Research Institute (KEMRI). The study will not recruit subjects prior to approval from both the University of Washington IRB and the KEMRI ERC.
   * Risks:

   Patients will be informed of all potential risks. The proposed study will involve adult men and women infected with HIV-1. All participants will be interviewed. Participants may experience discomfort while answering some of the questions regarding socio-economic status. Participants may also be uncomfortable discussing or providing stool samples for helminth screening. Study staff including social workers and/or peer counselors may contact the participants by telephone or visit the participants in their home if scheduled appointments are missed. These visits will be conducted in a manner designed to protect confidentiality but it is impossible to completely eliminate the risk of further social stigmatization for participants.

   This study involves serial blood specimen collection at 5 time points over a two year period (enrollment and months 6, 12, 18, and 24). The collection of these samples involves venipuncture which may cause discomfort, pain or bruising. Precautions will be taken to avoid bleeding by immediate application of a pack and pressure at the injection sites.

   All participants will provide written informed consent prior to screening or enrollment. Any adverse events associated with anti-helminthic medications will be managed by the appropriate clinic site, and if necessary, hospitalization. The costs of this care will be borne by the study. All clinical information including HIV status that is collected for the purposes of the study will be delinked from any client's identifier. This includes data collected in the clinic and in the laboratory. All data will be entered into a password protected computer with no links to identifiers. The code linking individual patient identifiers to a unique study ID will be kept securely locked in a separate location under control of the study principal investigator. All study files will be accessible only to researchers and will be stored in a locked office when not in use.

   There may be risks associated with use of the study medications, albendazole and praziquantel:

   Albendazole is a benzimidazole carbamate derivative with activity against most nematodes and some other worms. Albendazole is thought to inhibit cytoplasmic microtubules in the worm's intestinal tract leading to decreased glucose uptake and depletion of glycogen stores in the worm. Three 400 mg doses of albendazole has efficacy against whipworm, hookworm and roundworm infections, all of which we expect to be prevalent in this cohort. A recent randomized controlled trial of various albendazole dosing regimens showed that a single 400mg dose of albendazole was associated with a significantly lower rate of cure (23%) compared to a three day regimen (67%). In this study, reduction in the number of eggs/gm of feces with a single 400mg dose was 96.8% compared to 99.7% with the three day regimen. Albendazole is minimally absorbed from the gastrointestinal tract and has minimal side-effects.

   Praziquantel is a heterocyclic prazino-isoquinoline derivative with significant activity against both cestodes and trematodes. Praziquantel is highly effective against schistosomes in humans and there have been no confirmed cases of resistance reported. Praziquantel is well tolerated and severe adverse reactions are rare. There have been rare cases of increased intracranial pressure during treatment in patients with neurocysticercosis. This is not anticipated to be an issue in Kenya due to the low level of pork consumption in this population and the rarity of Taenia solium. In the study described above, we screened over 1600 individuals for helminths and documented no cases of Taenia solium (Walson J, unpublished data). Praziquantel is contraindicated in pregnancy and all female patients will undergo urine beta-HCG testing prior to administration. Pregnant or breast feeding women will not receive praziquantel.

   Patients with obvious clinical signs or symptoms of anaemia, significant diarrhoea or abdominal pain will not be enrolled. Neither routine screening of asymptomatic helminth infection nor empiric anti-helminth therapy is currently conducted in adults in Kenya.

   • Confidentiality: Patients will be assigned a study number at enrollment. This number will be used to identify patients for all matters related to data analysis. The forms linking patient names and demographic information to particular ID numbers will be kept locked in a file at the office of the Fellow Investigator.

   • Expected application of result: We anticipate that the proposed study will help to determine the role that common helminth co-infections play in HIV-1 pathogenesis and progression. If empiric deworming is found to significantly slow HIV-1 disease progression, it may be a cost-effective and easily implemented strategy to add to the current treatment options in helminth endemic areas.

ELIGIBILITY:
Inclusion Criteria:

* Participants must not be or have been on highly active antiretroviral therapy.
* Participants must have CD4 count > 350 cells/mm3 in order to be enrolled in the randomized controlled trial.
* Participants must be at least 18 years of age.
* Participants must be able and willing to participate and give written informed consent.
* Participants must be able and willing to return for the scheduled follow-up visits.

Exclusion Criteria:

• Participants must not be pregnant at the time of enrollment (by urine HCG testing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 948 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
CD4 count | every 6 months for 24 months (enrollment and months 6, 12, 18, and 24 )
  The primary measure of efficacy for the randomized clinical trial is the time to ART eligibility and the time to CD4 counts of less than 200 and 350 cells/mm3.
HIV-1 RNA level | enrollment, 12, and 24 months.

SECONDARY OUTCOMES:
Markers of clinical disease progression as measured by WHO staging criteria | Every 3 months for 24 months (enrollment, months 3, 6, 9, 12, 15, 18, 21, and 24)
  Secondary measures of efficacy will include changes in WHO Clinical Staging, development of IRIS, time to hospitalization, time to death, time to initiation of ARVs and CD4 response to ARVs as well as the development of IRIS among those who initiate ARVs.

CONTACTS AND LOCATIONS:
Overall Officials: Judd L Walson, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

REFERENCES:
- [Background] Fincham JE, Markus MB, Adams VJ. Could control of soil-transmitted helminthic infection influence the HIV/AIDS pandemic. Acta Trop. 2003 May;86(2-3):315-33. doi: 10.1016/s0001-706x(03)00063-9. PMID 12745148
- [Background] Bentwich Z, Weisman Z, Moroz C, Bar-Yehuda S, Kalinkovich A. Immune dysregulation in Ethiopian immigrants in Israel: relevance to helminth infections? Clin Exp Immunol. 1996 Feb;103(2):239-43. doi: 10.1046/j.1365-2249.1996.d01-612.x. PMID 8565306
- [Background] Kassu A, Tsegaye A, Wolday D, Petros B, Aklilu M, Sanders EJ, Fontanet AL, Van Baarle D, Hamann D, De Wit TF. Role of incidental and/or cured intestinal parasitic infections on profile of CD4+ and CD8+ T cell subsets and activation status in HIV-1 infected and uninfected adult Ethiopians. Clin Exp Immunol. 2003 Apr;132(1):113-9. doi: 10.1046/j.1365-2249.2003.02106.x. PMID 12653845
- [Background] Wolday D, Mayaan S, Mariam ZG, Berhe N, Seboxa T, Britton S, Galai N, Landay A, Bentwich Z. Treatment of intestinal worms is associated with decreased HIV plasma viral load. J Acquir Immune Defic Syndr. 2002 Sep 1;31(1):56-62. doi: 10.1097/00126334-200209010-00008. PMID 12352151
- [Background] Lawn SD, Karanja DM, Mwinzia P, Andove J, Colley DG, Folks TM, Secor WE. The effect of treatment of schistosomiasis on blood plasma HIV-1 RNA concentration in coinfected individuals. AIDS. 2000 Nov 10;14(16):2437-43. doi: 10.1097/00002030-200011100-00004. PMID 11101053
- [Derived] Means AR, van Lieshout L, Brienen E, Yuhas K, Hughes JP, Ndungu P, Singa B, Walson JL. Combined effectiveness of anthelmintic chemotherapy and WASH among HIV-infected adults. PLoS Negl Trop Dis. 2018 Jan 18;12(1):e0005955. doi: 10.1371/journal.pntd.0005955. eCollection 2018 Jan. PMID 29346385
- [Derived] Gerns Storey HL, Richardson BA, Singa B, Naulikha J, Prindle VC, Diaz-Ochoa VE, Felgner PL, Camerini D, Horton H, John-Stewart G, Walson JL. Use of principal components analysis and protein microarray to explore the association of HIV-1-specific IgG responses with disease progression. AIDS Res Hum Retroviruses. 2014 Jan;30(1):37-44. doi: 10.1089/AID.2013.0088. Epub 2013 Dec 9. PMID 24134221
- [Derived] Walson J, Singa B, Sangare L, Naulikha J, Piper B, Richardson B, Otieno PA, Mbogo LW, Berkley JA, John-Stewart G. Empiric deworming to delay HIV disease progression in adults with HIV who are ineligible for initiation of antiretroviral treatment (the HEAT study): a multi-site, randomised trial. Lancet Infect Dis. 2012 Dec;12(12):925-32. doi: 10.1016/S1473-3099(12)70207-4. Epub 2012 Sep 10. PMID 22971323